CLINICAL TRIAL: NCT04828278
Title: Effects of nooLVL Ingestion on Reaction Time and Cognitive Function in Gamers
Brief Title: Nutrition21 Study 1
Acronym: N21-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Nutrition 21, Inc. (Industry)
Responsible Party: Principal Investigator, Richard B. Kreider, Executive Director, Human Clinical Research Facility, Texas A&M University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB2020-0181D
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Nutritional Supplementation
MeSH Terms: interventions — Arginine

STUDY DESIGN:
Intervention Model Description: Crossover Intervention Trial
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment 1 (Placebo Comparator): 1,600 mg of Placebo (maltodextrin)
  Interventions: Dietary Supplement: Placebo
- Treatment 2 (Active Comparator): 1,500 mg of ASI (bonded arginine silicate) + 100 mg of inositol (nooLVL)
  Interventions: Dietary Supplement: Arginine

INTERVENTIONS:
Dietary Supplement: Arginine — Bonded Arginine Silicate
  Arms: Treatment 2
Dietary Supplement: Placebo — Maltodextrin
  Arms: Treatment 1

SUMMARY:
The purpose of this study is to determine the effects of nooLVL containing arginine and inositol supplementation on executive function and memory prior to and following playing video games.

DETAILED DESCRIPTION:
Gaming or "E-Sports" has become a very popular activity particularly among younger individuals. It requires quick reactions, executive function, memory and fine motor skill. In E-Sport competitions and tournaments, E-Sport players often play for hours per session over a series of days. Thus, the ability to maintain cognitive and executive function, concentration and fine motor skill is paramount. Two recent studies have evaluated the effects of ingesting bonded arginine silicate (ASI) and ASI with additional inositol on cognitive function. In the first study, ASI supplementation (1,500 mg/d for 3 days and 14 days) significantly improved the ability to perform complex cognitive tests requiring mental flexibility, processing speed and executive functioning. In the second study, adding 100 mg of inositol to the ASI significantly improved cognitive function in gamers after playing video games for one hour. This study is designed to assess the effects of bonded arginine silicate and inositol ingestion on reaction time and cognitive function prior to and following a 1-hour gaming challenge.

ELIGIBILITY:
Inclusion Criteria:

* They are a healthy male or female Gamer 18 to 40 years of age;
* They have a Body Mass Index (BMI) between 18 and 34.9 kg/m2;
* They are willing to supply their own operator-oriented action or stragegy video game that they have played 21 times over the last 3 months and the gaming platform with all accessories needed to play the chosen game;
* They report no recent ingestion (<2 weeks) of dietary supplements that affect cognitive function including nitrates and nitrous oxide (NO2) promoting supplements;
* They have a willingness to provide voluntary, written informed consent to participate in the study;

Exclusion Criteria:

* They have known cardiovascular, metabolic and/or other diseases under the treatment of a physician requiring prescription (Rx) medication (birth control is allowed);
* They have a history of cognitive dysfunction;
* They have a known allergy to maltodextrin;
* They have known allergies or asthma;
* They have cirrhosis;
* They have guanidinoacetate methyltransferase deficiency;
* They have herpes;
* They have abnormally low blood pressure;
* They have had a recent heart attack (i.e., within one year);
* They have kidney disease;
* They have a surgery scheduled in the next 4-5 weeks;
* Thye have had a gastrectomy;
* They have a bipolar disorder;
* They have an allergy to aspirin or tartrazine products;
* They are pregnant or breast-feeding or plan to become pregnant in the next 4-5 weeks;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Cognitive Function: Go No-Go Task Test | Measured prior to supplementation (Pre-Gaming), and after 15 and 60 minutes (Post-Gaming).
  General Attention Test
Cognitive Function: Phychomotor Vigilance Task Test | Measured prior to supplementation (Pre-Gaming), and after 15 and 60 minutes (Post-Gaming).
  Sustained Attention Test
Cognitive Function: Berg-Washington Card Sorting Task Test | Measured prior to supplementation (Pre-Gaming), and after 15 and 60 minutes (Post-Gaming).
  Attention Shifting Test
Cognitive Function: Sternberg Task Test | Measured prior to supplementation (Pre-Gaming), and after 15 and 60 minutes (Post-Gaming).
  Working Memory Test
Cognitive Function: Cambridge Brain Sciences Reasoning and Concentration Test | Measured prior to supplementation (Pre-Gaming), and after 15 and 60 minutes (Post-Gaming).
  Reasoning and Concentration Test
Cognitive Function: Light Tracking Reaction Time Test | Measured prior to supplementation (Pre-Gaming), and after 15 and 60 minutes (Post-Gaming).
  Reaction Time Test

SECONDARY OUTCOMES:
Gaming Score and Progression | Measured prior to supplementation (Pre) and after 60 minutes.
  Score and Progression
Stimulant Sensitivity Questionnaire | Measured prior to supplementation (Pre) and after 60 minutes.
  Stimulant Sensitivity
Side Effects Questionnaire | Measured prior to supplementation (Pre) and after 60 minutes.
  Side Effects

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Human Clinical Research Facility, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No